CLINICAL TRIAL: NCT03790111
Title: A Phase 2, Multicenter, Open-label, Safety and Efficacy Study of XERMELO® (Telotristat Ethyl) Plus First-line Chemotherapy in Patients With Locally Advanced, Unresectable, Recurrent or Metastatic Biliary Tract Cancer (BTC)
Brief Title: A Safety and Efficacy Study of XERMELO® + First-line Chemotherapy in Patients With Advanced Biliary Tract Cancer
Acronym: TELE-ABC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Did not meet pre-specified Progression-Free Survival at Month 6 for Stage 2 Analysis
Sponsor: TerSera Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LX1606.1-207-BTC; LX1606.207 (Other: TerSera Therapeutics); LX1606.207 (Other: Lexicon)
Record Dates: First submitted 2018-12-25; First posted 2018-12-31 (Actual); Results first posted 2023-04-19 (Actual); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Biliary Tract Cancer (BTC)
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — telotristat ethyl; Cisplatin; cytokine inducible SH2-containing protein

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Xermelo 250mg plus first line therapy for a week, then Xermelo 500mg (Experimental): Xermelo 250 milligram (mg) plus first line therapy for a week, then Xermelo 500mg plus first line therapy for the duration of the study
  Interventions: Drug: telotristat ethyl

INTERVENTIONS:
Drug: telotristat ethyl — XERMELO (telotristat ethyl) tablets administered as 250 mg (1 x 250-mg tablet) three times a day plus first line therapy for 7 days, then XERMELO (telotristat ethyl) tablets administered as 500 mg (2 x 250-mg tablets) three times a day plus first line therapy for the duration of the study
  Other Names: telotristat ethyl + (cisplatin [cis] plus gemcitabine [gem])

SUMMARY:
A Phase 2, multicenter, open-label, 2-stage study to assess the safety, tolerability, and efficacy of XERMELO in combination with first-line (1L) therapy (cisplatin [cis] plus gemcitabine [gem])

DETAILED DESCRIPTION:
A Phase 2, multicenter, open-label, 2-stage study to assess the safety, tolerability, and efficacy of XERMELO in combination with first-line (1L) therapy cis plus gem in patients with unresectable, locally advanced, recurrent or metastatic biliary tract cancer (intrahepatic or extrahepatic cholangiocarcinoma, gallbladder cancer), who are naïve to tumor-directed therapy in the locally advanced or metastatic setting, and for which treatment with 1L therapy (defined as a combination of cis plus gem) is planned.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults, ≥18 years of age. Patients of childbearing potential must agree to use an adequate method of contraception during the study and for 30 days after the last dose of XERMELO
* Histopathologically or cytologically-confirmed, unresectable, locally advanced, recurrent, or metastatic biliary tract cancer (BTC)
* Naïve to tumor-directed therapy in locally advanced, unresectable, or metastatic setting
* Measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Plans to initiate treatment with 1L therapy (cisplatin plus gemcitabine)
* Ability to provide written informed consent prior to participation in any study-related procedure

Exclusion Criteria:

* Prior exposure to XERMELO, telotristat ethyl, telotristat etiprate, LX1032, or LX1606
* Primary tumor site in the ampulla of Vater
* Treatment with photodynamic therapy for localized disease or to relieve biliary obstruction in the presence of metastatic disease within the past 30 days
* Hematology laboratory values of: a. Absolute neutrophil count (ANC) ≤1,500 cells/mm^3; or b. Platelets ≤100,000 cells/mm^3; or c. Hemoglobin (Hgb) ≤9 g/dL; or d. White blood count (WBC) ≤3,000 cells/mm^3
* Hepatic laboratory values of aspartate aminotransferase (AST) or alanine aminotransferase (ALT): a. >5 x upper limit of normal (ULN) if patient has documented history of hepatic metastases; or b. >2.5 x ULN if no liver metastases are present
* Serum albumin <2.8 g/dL
* Total bilirubin >1.5 x ULN or >1.5 mg/dL
* Prothrombin time (PT) or international normalized ratio (INR) >1.5 x ULN
* Serum creatinine or serum urea >1.5 x ULN
* Estimated glomerular filtration rate (eGFR) <50 mL/min
* Positive pregnancy test, pregnant, or breastfeeding
* Any other clinically significant laboratory abnormality that would compromise patient safety or the outcome of the study
* Any clinically significant and/or uncontrolled cardiac-related abnormality that would compromise patient safety or the outcome of the study
* Myocardial infarction within the past 6 months
* Active bleeding diathesis
* Life expectancy ≤3 months
* Current complaints of persistent constipation or history of chronic constipation, bowel obstruction or fecaloma within the past 6 months
* Receiving chronic treatment with corticosteroids ≥5 mg of prednisone per day (or equivalent) or other immunosuppressive agent(s)
* History and/or uncontrolled hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV Ab), or human immunodeficiency virus (HIV)-1 or HIV-2
* History of substance or alcohol abuse within the past 2 years
* History of galactose intolerance, deficiency of Lapp lactase, or glucose-galactose malabsorption
* History of malignancy or active treatment for malignancy within 5 years
* Receipt of live, attenuated vaccine or close contact with someone who has received a live, attenuated vaccine within the past 1 month
* Receipt of any investigational agent or study treatment (ie, any treatment or therapy not approved by the FDA for the treatment of BTC) within the past 30 days
* Receipt of any protein or antibody-based therapeutic agents within the past 3 months
* Treatment with any tumor-directed therapy within the past 6 months with curative intent
* Existence of any surgical or medical condition that, in the judgment of the Investigator, might compromise patient safety or the outcome of the study
* Presence of any clinically significant findings (relative to the patient population) during review of medical history or upon physical exam that, in the Investigator's or Medical Monitor's opinion, would compromise patient safety or the outcome of the study
* Evidence of brain metastases
* Unable or unwilling to communicate or cooperate with the Investigator for any reason
* Employee of Sponsor or clinical site, or relative of any member of a clinical site's staff

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2022-01-13 (Actual); Study Completion 2022-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Renuka Iyer, M.D., Study Chair — Roswell Park Cancer Institute; Richard Kim, M.D., Study Chair — H. Lee Moffitt Cancer Center and Research Institute
Locations (14):
- United States (14):
  - TerSera Investigational Site, Gilbert, Arizona
  - TerSera Investigational Site, Fullerton, California
  - TerSera Investigational Site, Gainesville, Florida
  - TerSera Investigational Site, Tampa, Florida
  - TerSera Investigational Site, Chicago, Illinois
  - TerSera Investigational Site, Westwood, Kansas
  - TerSera Investigational Site, Lexington, Kentucky
  - TerSera Investigational Site, Boston, Massachusetts
  - TerSera Investigational Site, Grand Rapids, Michigan
  - TerSera Investigational Site, Buffalo, New York
  - TerSera Investigational Site, Lake Success, New York
  - TerSera Investigational Site, Charlotte, North Carolina
  - TerSera Investigational Site, Oklahoma City, Oklahoma
  - TerSera Investigational Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg: Xermelo 250mg plus 1L therapy for a week, then Xermelo 500mg plus 1L therapy for the duration of the study
  telotristat ethyl: XERMELO (telotristat ethyl) tablets administered as 250 mg (1 x 250-mg tablet) tid plus 1L therapy for 7 days, then XERMELO (telotristat ethyl) tablets administered as 500 mg (2 x 250-mg tablets) tid plus 1L therapy for the duration of the study
Period: Overall Study
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Started | 53
Completed | 0 (Primary endpoint was not met. Study was early terminated.)
Not Completed | 53
Not completed — Study did not meet its primary endpoint. | 53

BASELINE CHARACTERISTICS:
Population: Safety Population
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.4 (10.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 46
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 53
Height [Mean (Standard Deviation); unit: inches] | 66.4 (3.37)
Weight [Mean (Standard Deviation); unit: kilogram] | 81.9 (17.40)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.85 (6.343)
Baseline Plasma 5-Hydroxyindoleacetic Acid (5-HIAA) Levels </= to ULN [Count of Participants; unit: Participants] — 5-HIAA: Normal (</=) was considered </= 10.8 micrograms/Liter High (>ULN) was considered >10.8 micrograms/Liter
  Participants
    </= ULN | 31
    >ULN | 22
Serum CA19-9 [Count of Participants; unit: Participants]
  Normal | 19
  Abnormal | 32
  Not Available | 2
Serum CEA [Count of Participants; unit: Participants]
  Normal | 25
  Abnormal | 26
  Not Available | 2
Serum Albumin [Count of Participants; unit: Participants]
  Normal | 48
  Abnormal | 4
  Not Available | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression-free Survival (PFS) as Evaluated by Central Radiologist's Assessment
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions", or similar definition as accurate and appropriate.
Time Frame: Month 6
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants
  Safety Population: Responders, Central Reviewer | 12
  Safety Population: Non-Responders, Central Reviewer | 41
  Per Protocol Population: number analyzed (Participants) | 42
  Per Protocol Population: Responders, Central Reviewer | 12
  Per Protocol Population: Non-Responders, Central Reviewer | 30
  By Treatment Cycle Population: number analyzed (Participants) | 33
  By Treatment Cycle Population: Responders, Central Reviewer | 12
  By Treatment Cycle Population: Non-Responders, Central Reviewer | 21

2. Primary Outcome: Project Overall Survival Rate at Month 6
Description: Overall Survival (OS) was defined as the time from the frist dose of study treatment until the date of death due to any cause. Duration of Overall Survival (OS) in days is defined as (Date of event/censoring- date of First dose +1). Use Kaplan Meier method to project survival rate at month 6.
Time Frame: 6 Months
Population: Safety Population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Proportion of participants | 0.87 [0.74 to 0.93]

3. Secondary Outcome: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the time from first dose of study treatment until the date of death due to any cause.
Time Frame: First dose of study treatment until the date of death due to any cause, whichever came first, a median of approximately 17.67 months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Months | 17.667 [11.567 to NA] — Due to insufficient number of participants with events, the upper margin cannot be estimated.

4. Secondary Outcome: Project Overall Survival Rate at Month 12
Description: Overall Survival (OS) was defined as the time from the first dose of study treatment until the date of death due to any cause. Duration of Overall Survival (OS) in days is defined as (Date of event/censoring - date of first dose +1). Use Kaplan Meier method to project survival rate at month 12.
Time Frame: 12 Months
Population: Safety population
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Proportion of participants | 0.60 [0.45 to 0.72]

5. Secondary Outcome: Median Progression Free Survival
Description: Scheduled disease assessment at Cycle 19 Day 1 was used to determine PFS response rate at Month 12.
Time Frame: Month 12
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Months | 6.233 [4.067 to 7.467]

6. Secondary Outcome: Disease Control Rate (DCR), Central Radiologist's Assessment
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.".
Time Frame: Month 6
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants | 33

7. Secondary Outcome: Disease Control Rate (DCR), Central Radiologist's Assessment
Description: Disease control rate (DCR) was defined as the proportion of patients with best overall response of SD longer than 6 weeks from first dosing, confirmed PR, or confirmed CR.
Time Frame: Month 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants | 33

8. Secondary Outcome: Disease Control Rate (DCR), Central Radiologist's Assessment
Description: as for outcome 7
Time Frame: End of Study up to 24 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants | 35

9. Secondary Outcome: Overall (Objective) Response Rate (ORR), Central Radiologist's Assessment
Description: Overall response rate (ORR) was defined as the proportion of patients with best overall response of confirmed PR or confirmed CR. The best overall response was the best overall response recorded from the start of study treatment until the EOS considering any requirement for confirmation.
  (CR) + partial response (PR) at Months 6
Time Frame: Month 6
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants | 7

10. Secondary Outcome: Overall (Objective) Response Rate (ORR), Central Radiologist's Assessment
Description: Overall response rate (ORR) was defined as the proportion of patients (Number of Responders) with best overall response of confirmed PR or confirmed CR. The best overall response was the best overall response recorded from the start of study treatment until Month 12.
Time Frame: Month 12
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants | 7

11. Secondary Outcome: Overall (Objective) Response Rate, Central Radiologist's Assessment
Description: Overall response rate (ORR) was defined as the proportion of patients with best overall response of confirmed PR or confirmed CR. The best overall response was the best overall response recorded from the start of study treatment until the EOS considering any requirement for confirmation.
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Participants | 7

12. Secondary Outcome: Summary of Duration of Progression Free Survival, Local Radiologist's Assessment
Description: Summary of Duration of Median Progression Free Survival, Local Radiologist's Assessment. Patient progression was defined from date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 7 months.
Time Frame: up to 7 months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Months | 7.000 [5.567 to NA] — Due to insufficient number of participants with events, the upper margin cannot be estimated.

13. Secondary Outcome: Progression Free Survival, Local Radiologist's Assessment
Description: Summary of Median Progression Free Survival, Local Radiologist's Assessment. Defined as the time from first dose of study treatment until the first date of either disease progression or death due to any cause. Scheduled disease assessment at Cycle 19 Day 1 was used to determine PFS response rate at Month 12.
Time Frame: Month 12
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Months | 7.467 [5.567 to 10.533]

14. Secondary Outcome: Progression Free Survival, Local Radiologist's Assessment
Description: Summary of Median Progression Free Survival, Local Radiologist's Assessment, End of Study
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 53
Months | 7.467 [5.567 to 10.533]

15. Secondary Outcome: Overall (Objective) Response Rate, Local Read
Description: Overall response rate (ORR) was defined as the proportion of patients with best overall response of confirmed PR or confirmed CR. The best overall response was the best overall response recorded from the start of study treatment at Month 6.
Time Frame: 6 Months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 48
Participants | 6

16. Secondary Outcome: Overall (Objective) Response Rate, Local Reader's Assessment
Description: Overall response rate (ORR) was defined as the proportion of patients with best overall response of confirmed PR or confirmed CR. The best overall response was the best overall response recorded from the start of study treatment at Month 12.
Time Frame: 12 Months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 48
Participants | 8

17. Secondary Outcome: Overall (Objective) Response Rate (ORR), Local Reader's Assessment
Description: as for outcome 11
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 48
Participants | 8

18. Secondary Outcome: Disease Control Rate (DCR), Local Reviewer
Description: as for outcome 7
Time Frame: Month 12 as defined by 1 year
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 48
Participants | 40

19. Secondary Outcome: Disease Control Rate (DCR), Local Reviewer
Description: Disease control rate (DCR), Local Reviewer, 6 Months
Time Frame: Month 6
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 48
Participants | 40

20. Secondary Outcome: Disease Control Rate End of Study, Local Reviewer
Description: as for outcome 7
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 48
Participants | 40

21. Secondary Outcome: Mean Change From Baseline in Plasma 5-hydroxyindoleacetic Acid (5-HIAA)
Description: Mean change from Baseline to Month 6 plasma level 5-hydroxyindoleacetic acid (5-HIAA)
Time Frame: Month 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micrograms/Liter
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 24
micrograms/Liter | -1.735 (8.6933)

22. Secondary Outcome: Mean Change From Baseline in Plasma 5-hydroxyindoleacetic Acid (5-HIAA)
Description: Mean change from Baseline to Month 12 in plasma level 5-hydroxyindoleacetic Acid (5-HIAA)
Time Frame: Month 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micrograms/Liter
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 6
micrograms/Liter | -5.608 (6.5192)

23. Secondary Outcome: Mean Change From Baseline in Plasma 5-hydroxyindoleacetic Acid (5-HIAA)
Description: Mean change from Baseline to End of Study in plasma 5-hydroxyindoleacetic acid (5-HIAA)
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: micrograms/Liter
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 7
micrograms/Liter | 4.154 (5.7003)

24. Secondary Outcome: Change From Baseline in Carbohydrate Antigen 19-9 (CA 19-9)
Description: Mean change from Baseline to month 6 in plasma carbohydrate antigen 19-9 (CA 19-9)
Time Frame: Month 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 21
U/mL | -229.82 (2484.902)

25. Secondary Outcome: Change From Baseline in Carbohydrate Antigen 19-9 (CA 19-9)
Description: Mean change from Baseline to Month 12 in plasma carbohydrate antigen 19-9 (CA 19-9)
Time Frame: Month 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 7
U/mL | -18.04 (38.665)

26. Secondary Outcome: Change From Baseline in Plasma Carbohydrate Antigen 19-9 (CA 19-9)
Description: Mean change from Baseline to End of Study in plasma carbohydrate antigen 19-9 (CA 19-9)
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Units per milliliter
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 8
Units per milliliter | -153.98 (456.210)

27. Secondary Outcome: Weight Change From Baseline
Description: Mean change in weight at Month 6 from baseline measurement
Time Frame: Month 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 17
kg | -0.69 (9.759)

28. Secondary Outcome: Weight Change From Baseline
Description: Mean change in weight at Month 12 from baseline measurement
Time Frame: Month 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 6
kg | 1.69 (7.473)

29. Secondary Outcome: Weight Change From Baseline
Description: Mean change in weight from baseline to End of Study
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 19
kg | -3.28 (8.920)

30. Secondary Outcome: Change From Baseline in Serum Albumin
Description: Mean change from Baseline to Month 6 serum albumin levels
Time Frame: Month 6
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 15
g/L | -0.2 (4.59)

31. Secondary Outcome: Change From Baseline in Serum Albumin
Description: Mean change from Baseline to Month 12 serum albumin levels
Time Frame: Month 12
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 6
g/L | -2.2 (2.86)

32. Secondary Outcome: Change From Baseline in Serum Albumin
Description: Mean change from Baseline to End of Study serum albumin levels
Time Frame: End of Study as defined up to 24 months
Population: Safety Population
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
Number analyzed (Participants) | 9
g/L | -1.2 (4.99)

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg
All-Cause Mortality (participants affected / at risk) | 3/53
Serious Adverse Events (participants affected / at risk) | 24/53
Other Adverse Events (participants affected / at risk) | 53/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg (N=53)
Gastrointestinal disorders (Gastrointestinal disorders) | 8 (8)
Infections and infestations (Infections and infestations) | 5 (5) — Bacteremia Klebsiella bacteremia Pneumonia Sepsis Septic shock Urinary tract infection
Hepatobiliary disorders (Hepatobiliary disorders) | 3 (3) — Cholangitis Hepatobiliary disease Hyperbilirubinemia
Nervous system disorders (Nervous system disorders) | 3 (3) — Cerebrovascular accident Embolic stroke
Cardiac Disorders (Cardiac disorders) | 2 (2) — Acute myocardial infarction Atrial fibrillation Cardiac arrest Myocardial infarction
Investigations (Investigations) | 2 (2) — Blood bilirubin increased
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1) — Anemia Leukocytosis
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1 (1) — Post procedural hematuria
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 1 (1) — Decreased appetite
Psychiatric disorders (Psychiatric disorders) | 1 (1) — Mental status changes
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1 (1) — Stevens-Johnson syndrome
Vascular disorders (Vascular disorders) | 1 (1) — Vena cava thrombosis
Respiratory, Thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 (5) — Pulmonary embolism Chronic obstructive pulmonary disease Pleural effusion
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Xermelo 250mg Plus 1L Therapy for a Week, Then Xermelo 500mg (N=53)
Constipation (Gastrointestinal disorders) | 34 (34)
Nausea (Gastrointestinal disorders) | 33 (33)
Fatigue (General disorders) | 32 (32)
Anemia (Blood and lymphatic system disorders) | 27 (27)
Neutrophil count decreased (Blood and lymphatic system disorders) | 22 (22)
Platelet count decreased (Blood and lymphatic system disorders) | 19 (19)
Diarrhea (Gastrointestinal disorders) | 18 (18)
Vomiting (Gastrointestinal disorders) | 17 (17)
White blood cell count decreased (Blood and lymphatic system disorders) | 14 (14)
Decreased appetite (Metabolism and nutrition disorders) | 13 (13)
Oedema peripheral (General disorders) | 12 (12)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Headache (Nervous system disorders) | 11 (11)
Hypertension (Vascular disorders) | 11 (11)
Pyrexia (General disorders) | 11 (11)
Abdominal pain (Gastrointestinal disorders) | 14 (14)

LIMITATIONS AND CAVEATS:
This study was halted prematurely as it did not meet pre-specified Progression-Free Survival at Month 6 for Stage 2 Analysis.

Due to early discontinuation of the study with limited data, the study results (data) at Month 12 and End of Study may be unreliable and uninterpretable.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-11-23): https://cdn.clinicaltrials.gov/large-docs/11/NCT03790111/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-03): https://cdn.clinicaltrials.gov/large-docs/11/NCT03790111/SAP_001.pdf